CLINICAL TRIAL: NCT06406881
Title: Combine Effect of Myofascial Release Technique and Ocular Muscle Exercise in Myopia With Eye Strain Headache Among University Students
Brief Title: Combine Effect Of Myofascial Release Technique and Ocular Muscle Exercise Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/01796
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Physical Therapy Modalities; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual therapy (Active Comparator): ocular muscle exercise like palm , blinking and pencil pushups neck isometric exercise
  Interventions: Other: physical therapy
- myofascial release therapy (Experimental): myofascial release technique along with ocular and neck isometric exercise.
  Interventions: Other: physical therapy; Other: myofascial release therapy

INTERVENTIONS:
Other: physical therapy — Ocular muscle exercise which is consist of three exercise like palm exercise, blinking exercise, pencil pushup exercise.
  3 sets of 10 repetition 5 days a week. As well as strengthening exercise the neck isometric exercise. each exercise consist of 3 sets of 5 repetition 5 days a week.
  Total of three sessions .
Other: myofascial release therapy — Experimental group given MFR along with neck isometric and ocular muscle exercise.
  myofascial release technique on sternocleidomastoid muscle and upper trapezius muscles. Patients will be treated 3 seconds to 2 minutes, three days in a week.
  Ocular muscle exercise will perform 3 sets of 10 repetition 5 days a week. As well as strengthening exercise the neck isometric exercise. This exercise will performed 3 sets of 5 repetition 5 days a week.
  Total of three sessions .
  Arms: myofascial release therapy

SUMMARY:
The current study aim to determine the effect of myofascial release technique and ocular muscle exercise to release eye strain headache in myopic students.

This study aim to reduce eye strain headache to improve quality of life and student academic performance. This study will enable the students to to work on digital device for a long period of time without any discomfort.

DETAILED DESCRIPTION:
According to recent researches MFR technique used to relax the muscles tension in muscles and fascia. This technique also enhance ROM. In this technique Apply gentle and sustain pressure on muscle start with light pressure gradually increase as it tolerated move the fingers along the length of muscle during apply pressure to take deep breath to help relax and facilitate the release.

Previous study showed a significant improvement in reduction of the number of headache days (p < 0.001) and the headache pain level (p < 0.001) following treatment.

The other intervention of this study is the ocular muscle exercise. Previous study showed that strengthening neck exercises like isometric neck exercise improve muscular strength and it is also delivering long term treatment effect on cervical pain.

This study divide in to two groups. Group A (experimental group) and Group B (control group)Patient in group A will receive ocular muscle exercise which is consist of three exercise like palm exercise, blinking exercise, pencil pushup exercise This group will also receive myofascial release technique on sternocleidomastoid muscle and upper trapezius muscles. Patient in group B will receive ocular muscle exercise and neck isometric exercise.

This study will manage the musculoskeletal and visual aspects of headaches and eye strain by combining myofascial release treatments with eye exercises. This study will contribute to reduce the eye strain headache and improve their quality of life and improve students' academic performance during class room and online learning.

ELIGIBILITY:
Inclusion Criteria:

* Age = 20- 30 years old
* Gender= male / female
* Diagnosed of Mild (-0.50 to -3.0 D) and moderate ( -3.0 to -6.0 D) myopia
* Unilateral or bilateral headache with mild or medium intensity
* Pain around eyes, forehead and temples
* Headache with neck stiffness or pain
* Headache increase with visual activity such as reading, using computer or cell phone.
* Headache associate with triggers in sternocleidomastoid, upper trapezius
* Positive convergent test (13)

Exclusion Criteria:

* History of genetic disease
* History of refractive surgery
* Wear contact lenses
* Headache associate with photophobia
* Headache associate with phonophobia
* History of neck trauma
* Cervical radiculopathy, herniated disc, arthritis
* Pain aggravated by movements of head

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Computer vision syndrome questionnaire | 5 days
  CVS is consist of 13 sections its scoring in the form of mild, moderate severe,

SECONDARY OUTCOMES:
tape measure method | 5 days
  Tape used to measure the length of muscle ( SCM, upper trapezius ) measurement from the baseline to third week.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Ghias, MS, Principal Investigator — Riphah International University
Locations (1):
- Abasyn university peshawar, Peshawar, Khyber Pakhtunkhawa, Pakistan

IPD SHARING:
Plan to Share IPD: No